CLINICAL TRIAL: NCT04015856
Title: Impact Evaluation of the Tipping Point Project in Nepal: An Intervention to Prevent Early Child Marriage
Brief Title: Preventing Early Child Marriage in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Cooperative for Assistance and Relief Everywhere, Inc. (CARE) (Unknown)
Responsible Party: Principal Investigator, Kathryn Yount, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00109419
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Child Marriage
Keywords: Social research

STUDY DESIGN:
Intervention Model Description: Wards (the lowest government administrative units in Nepal) will be treated as clusters or the primary sampling units in this study. Each cluster will be randomly assigned to one of the three arms. Adolescents residing in the study wards will be recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full TP intervention including emphasized social norms change (Experimental): Participants in this study arm will receive the full TP intervention, including emphasized social norms change, for 18 months.
  Interventions: Behavioral: Full TP intervention
- Light TP intervention without emphasized social norms change (Active Comparator): Participants in this study arm will receive the light TP intervention, without emphasized social norms change, for 18 months
  Interventions: Behavioral: Light TP intervention
- Control (No Intervention): The control group will not have any study interventions.

INTERVENTIONS:
Behavioral: Full TP intervention — CARE's Tipping Point initiative focuses on addressing the root causes of child, early, and forced marriage (CEFM) and promoting the rights of adolescent girls through community-level programming and evidence generation in Nepal and Bangladesh, as well as multi-level advocacy and cross-learning efforts across the globe. Tipping Point's approach focuses on synchronized engagement with different participant groups-including adolescent girls, adolescent boys, parents/community members, community leaders-around key programmatic pillars, and creates public spaces for all community members to engage in the dialogue. Tipping Point's approach relies on challenging social expectations and repressive gender norms and promoting girl-centric and girl-led activism to enable adolescent girls to identify and move into social spaces where they can challenge inequality.
  Arms: Full TP intervention including emphasized social norms change
Behavioral: Light TP intervention — The Tipping Point project also has designed a social norms light package, which includes a subset of the social norms and activism components of the full package.
  Arms: Light TP intervention without emphasized social norms change

SUMMARY:
This project evaluates an intervention designed to prevent early child marriage in Nepal. The intervention consists of community dialogues, activist trainings, and community organized activities aimed at transforming social norms around gender. There will be three groups within the study: one exposed to the full program, one exposed to a lighter version of the program, and one that has not been exposed to the program. The impact evaluation will consist of qualitative and quantitative methods that compare these three groups.

DETAILED DESCRIPTION:
Each year, child marriage, before age 18 years, affects more than 10 million girls globally. The practice is associated with adverse maternal and child health outcomes and diminished long-term economic empowerment. About half of all child marriages occur in South Asia. A recent study in four high prevalence South Asian countries showed declines in girl-child marriage from 1991-1994 to 2005-2007, however, these declines were concentrated in the youngest ages. Namely, significant relative reductions occurred in the marriage of girls before age 14 years in all countries, however, little or no change was seen in the marriage of 16- to 17-year-old girls for any country except Bangladesh, where the prevalence of such marriages increased.

Tipping Point (TP) is an innovative program developed by Cooperative for Assistance and Relief Everywhere, Inc. (CARE) to change community social norms and build capacity among adolescent girls to become agents of change in their communities, with the ultimate goal of reducing the risk of child marriage.

The quantitative evaluation of the TP package will involve a three arm Cluster Randomized Controlled Trial (CRCT), where the arms are as follows:

* Arm 1: Full TP intervention including emphasized social norms change
* Arm 2: Light TP intervention without emphasized social norms change
* Arm 3: Pure control

The overall evaluation in Nepal will start with the baseline study, followed by eighteen months of interventions. After the intervention phase, there will be a one year 'freeze' period, when no interventions will take place. After that one year, the end-line evaluation study will be conducted in Nepal to assess the impact of the packages.

ELIGIBILITY:
Inclusion Criteria for Clusters

* marginalized communities based on CARE Nepal formula
* communities prioritized by Nepal Government
* no concurrent non-governmental organization (NGO) programming
* no concurrent CARE programming

Inclusion Criteria for Boys and Girls (invited to participate in the intervention, survey, in-depth interviews, focus group discussions)

* unmarried
* age 12 -under 17
* living in study community
* no plans to migrate in subsequent 24 months

Inclusion Criteria for Mothers and Fathers of Selected Boys and Girls (invited to intervention and focus group discussions)

* male and female parental figures of an adolescent who has been recruited to participate in the intervention and associated measurement

Exclusion Criteria for Mothers and Fathers of Selected Boys and Girls:

* none

Inclusion Criteria for Community Adults:

* at least 25 years of age
* living in one of the study Communities
* no plans to migrate during the next two years

Exclusion Criteria for Community Adults:

* none

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2828 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Change in proportion of never married adolescents | Baseline, Month 30
  The proportion of never-married adolescents (aged under 20) in each study arm will be examined.
Change in proportion of married adolescents | Baseline, Month 30
  The proportion of married adolescents (aged under 20) in each study arm will be examined.

SECONDARY OUTCOMES:
Change in decision making | Baseline, Month 30
  Qualitative questions on gender and rights will assess awareness of rights, progressive choices, negotiation skills, and decision making of adolescent girls. Information will be collected during interviews asking open ended questions.
Change in Adolescent Sexual and Reproductive Health and Rights (ASRHR) | Baseline, Month 30
  Qualitative questions on ASRHR will assess the knowledge, progressive attitudes and practice of sexual and reproductive health rights among adolescent girls. Information will be collected during interviews asking open ended questions.
Change in social norms | Baseline, Month 30
  Qualitative questions on social norms change will assess to what extent the beliefs have shifted in the community regarding what others do in terms of gender, rights (including ASRHR) and child, early and forced marriage (CEFM) and what others expect them to do in terms of gender, rights (including ASRHR) and CEFM. Information will be collected during interviews asking open ended questions.
Change in movement building among adolescent girls | Baseline, Month 30
  Qualitative questions on girl-centered movement building will assess the cohesion, solidarity, leadership and mobilization skills of adolescent girls, as well as the adolescent girls' autonomous engagement with different networks, the community and government and non-government stakeholders. Information will be collected during interviews asking open ended questions.
Change in gender attitudes among community adults | Baseline, Month 30
  Adults in the intervention communities will complete a 42-item questionnaire about gender attitudes. The instrument includes the domains of gender roles, roles of girls and women, manhood and masculinity, controlling behaviors, and attitudes condoning violence against girls. Responses are given on a scale from 1 to 4 where 1 = fully agree and 4 = fully disagree. Summed scores range from 42 to 168, where higher scores indicate greater change in social norms.
Change in attitudes on ASRHR among community adults | Baseline, Month 30
  Adults in the intervention communities will complete a 16-item questionnaire about ASRHR attitudes. Responses are given on a scale from 1 to 4 where 1 = fully agree and 4 = fully disagree. Summed scores range from 16 to 64, where higher scores indicate greater change in social norms.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Yount, PhD, Principal Investigator — Emory University
Locations (1):
- Interdisciplinary Analysts, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Full baseline and endline datasets will be made available for sharing.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data will be available for sharing upon acceptance of main results for publication or 24 months after completion of endline, whichever comes first.
Access Criteria: Individual participant data will be accessible by written permission of the project principal investigators for analyses not related to the primary aims of this study, unless to test reproducibility. Access to the data can be requested by writing to the CARE Tipping Point Program Director anne.sprinkel@care.org

REFERENCES:
- [Derived] Clark CJ, Jashinsky K, Renz E, Bergenfeld I, Durr RL, Cheong YF, Kalra S, Laterra A, Yount KM. Qualitative endline results of the tipping point project to prevent child, early and forced marriage in Nepal. Glob Public Health. 2023 Jan;18(1):2287606. doi: 10.1080/17441692.2023.2287606. Epub 2023 Dec 6. PMID 38054604
- [Derived] Yount KM, Durr RL, Bergenfeld I, Sharma S, Clark CJ, Laterra A, Kalra S, Sprinkel A, Cheong YF. Impact of the CARE Tipping Point Program in Nepal on adolescent girls' agency and risk of child, early, or forced marriage: Results from a cluster-randomized controlled trial. SSM Popul Health. 2023 Apr 17;22:101407. doi: 10.1016/j.ssmph.2023.101407. eCollection 2023 Jun. PMID 37251506
- [Derived] Yount KM, Clark CJ, Bergenfeld I, Khan Z, Cheong YF, Kalra S, Sharma S, Ghimire S, Naved RT, Parvin K, Al Mamun M, Talukder A, Laterra A, Sprinkel A; Tipping Point Program Study Team. Impact evaluation of the Care Tipping Point Initiative in Nepal: study protocol for a mixed-methods cluster randomised controlled trial. BMJ Open. 2021 Jul 26;11(7):e042032. doi: 10.1136/bmjopen-2020-042032. PMID 34312191